CLINICAL TRIAL: NCT06376058
Title: Intrathecal Use of Chloroprocaine 1% and Ropivacaine 0,75% During Elective Cesarean Section. A Comparative Study
Brief Title: Chloroprocaine 1% Versus Ropivacaine 0,75% During Cesarean Section
Acronym: annie-mariana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 434/06-06-2022
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section; Local Anesthetic
MeSH Terms: interventions — chloroprocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chloroprocaine group (Active Comparator): intrathecal fixed dose of chloroprocaine 1%
  Interventions: Drug: Chloroprocaine 1% Injectable Solution
- ropivacaine group (Active Comparator): intrathecal fixed dose of ropivacaine 0.75%
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution

INTERVENTIONS:
Drug: Chloroprocaine 1% Injectable Solution — • in parturients allocated to the chloroprocaine group, a fixed dose of chloroprocaine 1% will be administered intrathecally
  Arms: chloroprocaine group
Drug: Ropivacaine 0.75% Injectable Solution — • in parturients allocated to the ropivacaine group, a fixed dose of ropivacaine 0.75% will be administered intrathecally
  Arms: ropivacaine group

SUMMARY:
This will be a prospective randomized study, aiming at comparing an intrathecal fixed dose of chloroprocaine 1% versus an intrathecal fixed dose of ropivacaine 0.75% in elective cesarean sections

DETAILED DESCRIPTION:
Neuraxial techniques are the anesthetic techniques of choice in contemporary obstetric anesthesia practice, with a definitive superiority as compared to general anesthesia, since, by their use, serious complications involving the airway can be avoided. Combined spinal-epidural anesthesia has become the favorable technique for both elective and emergency cesarean sections. Various local anesthetics have been used, but ropivacaine is the drug of choice in most hospitals in Greece. However, chloroprocaine is a preferable local anesthetic in USA due to its quick and predictable onset of action. Chloroprocaine was initially used in 1980, but it became obsolete in those years due to neurological symptoms associated with its use caused mainly by the presence of sodium bisulfite and disodium ethylenediaminetetraacetate (EDTA) in the early formulations. Nowadays, new formulations of the drug without EDTA makes chloroprocaine safe for use.

The aim of the current randomized controlled trial will be to compare the effect of an intrathecal fixed dose of chloroprocaine versus an intrathecal fixed dose of ropivacaine in parturients subjected to elective cesarean section under combined spinal-epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* adult parturients, American Society of Anesthesiologists (ASA) I-II,
* singleton gestation>37 weeks
* elective cesarean section

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) > III
* age < 18 years
* singleton gestation <37 weeks
* Body Mass Index (BMI) >40 kg/m2
* Body weight <50 kg
* Body weight>100 kg
* height<150 cm
* height>180 cm
* multiple gestation
* emergency delivery
* fetal abnormality
* fetal distress
* pregnancy-induced pathology such as preeclampsia, eclampsia, premature labor, placental abnormalities
* pregnancy- induced diseases such as hepatic failure, pseudocholinesterase deficiency, neuromuscular diseases
* lack of informed consent
* contraindication for regional anesthesia such as thrombocytopenia, coagulation abnormalities, allergy to local anesthetics

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Time from spinal anesthesia to T10 block (min) | intraoperative
  time required from spinal anesthetic injection to anesthetic block up to the 10th thoracic neurotome
Time from spinal anesthesia to T4 block (min) | intraoperative
  time required from spinal anesthetic injection to anesthetic block up to the 4th thoracic neurotome
Time of spinal anesthesia to Bromage =3 | intraoperative
  time required from spinal anesthetic injection to complete motor block (Bromage scale=3, where Bromage=0, no block; Bromage=1, partial block; Bromage=2, almost complete block; Bromage=3, complete block
level of sensory block every 3 min | intraoperative
  measurement of sensory block every 3 minutes after spinal anesthesia during the first 15 minutes
level of sensory block every 15 min | intraoperative
  measurement of sensory block every 15 minutes from spinal anesthesia to the end of the surgery
highest level of sensory block | intraoperative
  measurement of the highest level of sensory block after intrathecal infusion of local anesthetic
time from spinal anesthesia to highest level of sensory block | intraoperative
  time from the performance of spinal anesthesia to the highest level of sensory block
duration of sensory block | intraoperative
  measurement of time required for the sensory block to regress from sensory level T4 to sensory level T12/L2
pain at surgical incision | intraoperative
  pain at skin incision using Visual Analogue Scale (VAS), where VAS=0, no pain; VAS=10, worst pain imaginable
pain at neonatal delivery | intraoperative
  pain at neonatal delivery using VAS scale, where VAS=0, no pain; VAS=10, worst pain imaginable
pain at peritoneal manipulation | intraoperative
  pain at peritoneal manipulation using VAS scale, where VAS=0, no pain; VAS=10, worst pain imaginable
pain at Post Anesthesia Care Unit (PACU) admission | 1 hour postoperatively
  pain at Post Anesthesia Care Unit (PACU) admission using VAS scale, where VAS=0, no pain; VAS=10, worst pain imaginable
pain at Post Anesthesia Care Unit (PACU) discharge | 1 hour postoperatively
  pain at Post Anesthesia Care Unit (PACU) discharge using VAS scale, where VAS=0, no pain; VAS=10, worst pain imaginable
need for rescue analgesia intraoperatively | intraoperative
  need for rescue analgesia during the operation, via epidural catheter or intravenously
Bromage scale every 3 min after spinal anesthesia | intraoperative
  measurement of bromage scale every 3 minutes after spinal anesthesia during the first 15 minutes
Bromage scale every 15 min | intraoperative
  measurement of bromage scale every 15 minutes from spinal anesthesia to the end of the surgery
duration of motor block | 1 hour postoperatively
  measurement of time required for bromage scale to regress from 3 to 0
duration of staying in PACU | 2 hours postoperatively
  duration of parturient stay in PACU

SECONDARY OUTCOMES:
Neonatal Apgar score at 1 minute | 1 minute post delivery
  Neonatal Apgar score will be recorded at 1 minute after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts
Neonatal Apgar score at 5 minutes | 1 minute post delivery
  Neonatal Apgar score will be recorded at 5 minutes after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts
neonatal blood gases | 1 minute post delivery
  fetal cord blood analysis will be performed immediately post-delivery
incidence of neonatal acidosis | 1 minute post delivery
  incidence of neonatal acidosis (PH<7.2) will be recorded
incidence of hypotension | intraoperative
  any occurence of hypotension (systolic blood pressure<80% of baseline) throughout the operation will be recorded
incidence of bradycardia | intraoperative
  any incidence of maternal bradycardia (heart rate<60/min) will be recorded
need for vasoconstrictor | intraoperative
  any need for vasoconstrictor during the operation will be recorded
need for atropine | intraoperative
  any need for atropine during the operation because of bradycardia will be recorded
incidence of nausea/vomiting | intraoperative
  any occurence of nausea and/or vomiting during the operation will be recorded
incidence of dizziness | intraoperative
  any occurence of dizziness during the operation will be recorded
incidence of drowsiness | intraoperative
  any occurence of drowsiness during the operation will be recorded
incidence of discomfort | intraoperative
  any occurence of discomfort during the operation will be recorded
incidence of shivering | intraoperative
  any occurence of shivering during the operation will be recorded
need for rescue analgesia in PACU | 2 hours postoperatively
  need for rescue analgesia in PACU when VAS scale >4 will be recorded
time from spinal anesthesia to rescue analgesia in PACU | 2 hours postoperatively
  time from spinal anesthesia to rescue analgesia in PACU will be recorded
incidence of neurological symptoms during hospital stay | 5 days postoperatively
  incidence of neurological symptoms during hospitalization will be recorded
incidence of neurological symptoms 2 months after the operation | 2 months after discharge
  incidence of neurological symptoms 2 months after discharge from the hospital will be recorded by phone communication
incidence of low back pain | 2 months after discharge
  incidence of low back pain 2 months after discharge from the hospital will be recorded by phone communication
time from spinal anesthesia to mobilization | 2 days postoperatively
  time from spinal anesthesia to mobilization of parturient will be recorded
mother's satisfaction from anesthesia | 1 day postoperatively
  mother's satisfaction from anesthesia will be recorded using Likert scale. Likert scale ranges from 1 which is the minimum satisfaction to 4 which is the maximum satisfaction
gynecologist's satisfaction | 1 hour postoperatively
  gynecologist's satisfaction from anesthesia will be recorded using Likert scale. Likert scale ranges from 1 which is the minimum satisfaction to 4 which is the maximum satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Maes S, Laubach M, Poelaert J. Randomised controlled trial of spinal anaesthesia with bupivacaine or 2-chloroprocaine during caesarean section. Acta Anaesthesiol Scand. 2016 May;60(5):642-9. doi: 10.1111/aas.12665. Epub 2015 Nov 26. PMID 26608876
- [Background] Saporito A, Ceppi M, Perren A, La Regina D, Cafarotti S, Borgeat A, Aguirre J, Van De Velde M, Teunkens A. Does spinal chloroprocaine pharmacokinetic profile actually translate into a clinical advantage in terms of clinical outcomes when compared to low-dose spinal bupivacaine? A systematic review and meta-analysis. J Clin Anesth. 2019 Feb;52:99-104. doi: 10.1016/j.jclinane.2018.09.003. Epub 2018 Sep 18. PMID 30237085
- [Background] Singariya G, Choudhary K, Kamal M, Bihani P, Pahuja H, Saini P. Comparison of analgesic efficacy of intrathecal 1% 2-chloroprocaine with or without fentanyl in elective caesarean section: A prospective, double-blind, randomised study. Indian J Anaesth. 2021 Feb;65(2):102-107. doi: 10.4103/ija.IJA_816_20. Epub 2021 Feb 10. PMID 33776083
- [Background] Baribeault T, Suss S. Spinal Anesthesia with 2-Chloroprocaine and Dexmedetomidine for Cesarean Section: A Case Report. AANA J. 2023 Jun;91(3):194-196. PMID 37227957